CLINICAL TRIAL: NCT00096668
Title: A Phase 2 Multicenter Evaluation of the Safety and Efficacy of TOCOSOL(R) Paclitaxel (S-8184 Paclitaxel Injectable Emulsion) as Initial Treatment of Patients With Metastatic Breast Cancer
Brief Title: Evaluation of Safety and Efficacy of TOCOSOL(R) Paclitaxel as Initial Treatment for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Monica Krieger, VP Regulatory Affairs, OncoGenex Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SON-8184-1074
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; TOCOSOL Paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

ARMS (1):
- TOCOSOL Paclitaxel (Experimental): TOCOSOL Paclitaxel administered weekly at 120mg/mm2
  Interventions: Drug: TOCOSOL(R) Paclitaxel

INTERVENTIONS:
Drug: TOCOSOL(R) Paclitaxel

SUMMARY:
This is an open label study where each patient will receive TOCOSOL(R) Paclitaxel 120mg/m2 every week for first line treatment of metastatic breast cancer. Patients will be followed to determine the efficacy of treatment (as measured by objective response rate), and the safety associated with weekly administration of TOCOSOL Paclitaxel.

DETAILED DESCRIPTION:
This is an open label, non-randomized Phase 2 study of weekly administration of TOCOSOL Paclitaxel at a dose level, 120mg/m2, known to be tolerated based on Phase 2a studies of this investigational agent in patients with other histological diagnoses. This study is a fixed sample size design with no planned early stopping decision. The goals of the study include the determination of the safety of TOCOSOL Paclitaxel, and the objective response rate, defined by RECIST criteria as complete responses plus partial responses.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with histologic diagnosis of breast carcinoma
* Stage IV (M1) disease
* No prior cytotoxic chemotherapy regimen for treatment of metastatic breast cancer
* Adult (18 years of age or older) patients
* Adequate hematologic function (ANC >=1500 cells/mm3 and platelets >100,000/mm3
* Serum creatinine <=2.0 mg/dL
* Total bilirubin <=1.5 mg/dL
* AST/SGOT and ALT/SGPT <=3 times the upper limit of institutional normal values
* PT and PTT within institutional normal range
* ECOG performance status of 0-2
* At least one unidimensionally measurable lesion as defined by RECIST criteria assessable by radiographic evaluation
* A signed IRB/Ethics Committee approved Informed Consent
* Life expectancy of at least 12 weeks
* Fully recovered from any previous surgery
* A negative pregnancy test prior to study entry if premenopausal
* Agree not to take Vitamin E supplementation while receiving study medication

Exclusion Criteria:

* Any prior taxane-containing chemotherapy including Taxol or Taxotere
* Patients who are pregnant or lactating
* Peripheral neuropathy NCI-CTC grade 2 or greater
* Wide-field radiation, hormonal therapy or trastuzumab within 4 weeks of first dose of study drug; cytotoxic chemotherapy within 6 months of first dose of study drug
* Treatment with an investigational agent within 4 weeks of first dose of study drug
* Patients with a history of carcinomas of primary sites which can not be distinguished histologically from metastatic breast carcinoma
* Bone metastasis, effusions, ascites or elevated tumor markers as the only evidence of metastatic breast carcinoma
* Brain metastases
* Active bowel obstruction
* Active, serious infection or other serious medical problems (other than metastatic breast cancer) likely to impair completion of the study protocol
* Concurrent therapy with known substrates or inhibitors of the cytochrome P450 isoenzymes CYP2C8 or CYP3A4
* Concurrent therapy with warfarin or other coumarin derivatives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Tolerability | After all patients complete treatment

SECONDARY OUTCOMES:
Objective Response Rate | After alll patients complete treatment

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - Arkhangelsk Regional Oncology Center, Arkhangelsk
  - Moscow Oncology Clinical Hospital #62, Krasnogorskiy Region
  - Blokhin Russian Oncology Center, Moscow
  - Semashko Central Clinical Hospital of the Ministry of Transport, Moscow
  - St Petersburg Oncology Center, Saint Petersburg
  - Petrov Research Institute of Oncology, Saint Petersburg
  - Voronezh Regional Clinical Oncology Center, Voronezh